CLINICAL TRIAL: NCT01985334
Title: A Prospective, Multicenter, 12-week, Randomized Open-label Study to Evaluate the Efficacy and Safety of Glycopyrronium (50 Micrograms o.d.) or Indacaterol Maleate and Glycopyrronium Bromide Fixed-dose Combination (110/50 Micrograms o.d.) Regarding Symptoms and Health Status in Patients With Moderate Chronic Obstructive Pulmonary Disease (COPD) Switching From Treatment With Any Standard COPD Regimen
Brief Title: Study to Evaluate the Efficacy and Safety of Glycopyrronium or Indacaterol Maleate and Glycopyrronium Bromide Fixed-dose Combination Regarding Symptoms and Health Status in Patients With Moderate COPD Switching From Treatment With Any Standard COPD Regimen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQVA149A3401
Record Dates: First submitted 2013-11-04; First posted 2013-11-15 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: COPD
Keywords: Moderate COPD, glycopyrronium bromide, indacaterol maleate and glycopyrronium bromide FDC, NVA237, QVA149
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; 3-(2-(4-azidobenzamidino)ethyl)-5-hydroxyindole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- A1 (any SABA and/or SAMA) (Experimental): Patients treated with any SABA and/or SAMA as monotherapy or in free or fixed dose combination will be assigned to glycopyrronium or will remain in their baseline therapy (3:1) during 90 days of treatment
  Interventions: Drug: Glycopyrronium; Drug: SABA; Drug: SAMA
- A2 (glycopyrronium) (Experimental): Patients treated with any SABA and/or SAMA as monotherapy or in free or FDC at enrollment and randomized to switch in treatment with glycopyrronium (50 μg o.d.)
  Interventions: Drug: Glycopyrronium; Drug: SABA; Drug: LABA; Drug: SAMA
- B1 (any LAMA or LABA and mMRC=1) (Experimental): Patients treated with any LABA or LAMA monotherapy and mMRC score =1 point at Visit 1 and randomized to remain in their baseline treatment with LABA or LAMA
  Interventions: Drug: LABA; Drug: Indacaterol maleate and glycopyrronium bromide; Drug: LAMA; Drug: ICS
- B2 (glycopyrronium and mMRC=1) (Experimental): Patients treated with any LABA or LAMA monotherapy and mMRC score =1 point at Visit 1 and randomized to switch in treatment with glycopyrronium (50 μg o.d.)
  Interventions: Drug: LABA; Drug: Indacaterol maleate and glycopyrronium bromide; Drug: LAMA
- C1 (any LABA and ICS) (Experimental): Patients treated with any LABA and ICS in free or FDC at enrollment and randomized to remain in their baseline treatment with LABA and ICS in free or FDC
  Interventions: Drug: LABA; Drug: ICS
- C2 (indacaterol/glycopyrronium) (Experimental): Patients treated with any LABA and ICS in free or FDC at enrollment and randomized to switch in treatment with indacaterol maleate and glycopyrronium bromide FDC (110/50 μg o.d.)
  Interventions: Drug: LABA; Drug: ICS
- D1 (any LAMA or LABA and mMRC>1) (Experimental): Patients treated with any LABA or LAMA monotherapy and mMRC score >1 point at Visit 1 and randomized to remain their baseline in treatment with LABA or LAMA
  Interventions: Drug: LAMA
- D2 (indacaterol/glycopyrronium and mMRC>1) (Experimental): Patients treated with any LABA or LAMA monotherapy and mMRC score >1 point at Visit 1 and randomized to switch in treatment with indacaterol maleate and glycopyrronium bromide FDC (110/50 μg o.d.).
  Interventions: Drug: LAMA

INTERVENTIONS:
Drug: Glycopyrronium — Glycopyrronium 50 µg capsule for inhalation via SDDPI once per day
  Other Names: glycopyrronium bromide
  Arms: A1 (any SABA and/or SAMA); A2 (glycopyrronium)
Drug: SABA — Short-acting β2-adrenergic agonist (SABA) as per approved by each country and as prescribed for each patient, used as background therapy
  Arms: A1 (any SABA and/or SAMA); A2 (glycopyrronium)
Drug: LABA — Long Acting Beta Agonist (LABA) as per approved by each country and as prescribed for each patient, used as background therapy
  Arms: A2 (glycopyrronium); B1 (any LAMA or LABA and mMRC=1); B2 (glycopyrronium and mMRC=1); C1 (any LABA and ICS); C2 (indacaterol/glycopyrronium)
Drug: Indacaterol maleate and glycopyrronium bromide — Indacaterol maleate and glycopyrronium bromide fixed dose combination (110/50 µg) capsule for inhalation via SDDPI, once a day
  Arms: B1 (any LAMA or LABA and mMRC=1); B2 (glycopyrronium and mMRC=1)
Drug: LAMA — Long Acting Muscarinic Antagonist (LAMA) as per approved by each country and as prescribed for each patient, used as background therapy
  Arms: B1 (any LAMA or LABA and mMRC=1); B2 (glycopyrronium and mMRC=1); D1 (any LAMA or LABA and mMRC>1); D2 (indacaterol/glycopyrronium and mMRC>1)
Drug: SAMA — Short-acting muscarinic antagonist (SAMA) as per approved by each country and as prescribed for each patient, used as background therapy
  Arms: A1 (any SABA and/or SAMA); A2 (glycopyrronium)
Drug: ICS — Inhaled corticosteroid (ICS) as per approved by each country and as prescribed for each patient, used as background therapy
  Arms: B1 (any LAMA or LABA and mMRC=1); C1 (any LABA and ICS); C2 (indacaterol/glycopyrronium)

SUMMARY:
The main goal of this study is to evaluate the efficacy and safety of glycopyrronium bromide and indacaterol maleate and glycopyrronium bromide fixed dose combination (FDC) in patients with moderate COPD who switch from their current COPD therapy. This study aims to provide data on how non-exacerbating, but still symptomatic patients with moderate COPD switching from their current COPD treatment to glycopyrronium bromide or indacaterol maleate and glycopyrronium bromide FDC maintain or improve their symptoms. Another purpose of this study is to increase awareness and usage of validated COPD symptoms tools and dyspnea questionnaires in order to facilitate clinical assessment and improve early diagnosis of symptomatic patients.

DETAILED DESCRIPTION:
The treatment epoch will last 12 weeks. The total duration of the study for each patient is 12 weeks (from randomization) plus 30 days of safety follow-up.

The study has three phases: screening phase (=wash-out period, if required), treatment phase and safety follow-up phase.

Eligible patients will be randomized to either receive glycopyrronium or indacaterol maleate and glycopyrronium bromide fixed dose combination or to remain in their baseline therapy, in an allocation ratio of 3:1 for each cluster (Groups A, B, C, and D), based on their COPD symptoms and baseline treatment:

Group A: Patients treated with any SABA ( Short-acting β2-adrenergic agonist) and/or SAMA (Short-acting muscarinic antagonist) as monotherapy or in free or fixed dose combination (FDC) will be assigned to glycopyrronium or will remain in their baseline therapy (3:1) Group B: Patients treated with any LABA (Long-acting β2-adrenergic agonist) or LAMA (Long-acting muscarinic antagonist) monotherapy and mMRC score =1 point will be assigned to glycopyrronium or will remain in their baseline therapy (3:1) Group C: Patients treated with any LABA and ICS (Inhaled corticosteroid) in free or FDC will be assigned to indacaterol maleate and glycopyrronium bromide fixed dose combination or will remain in their baseline therapy (3:1) Group D: Patients treated with any LABA or LAMA monotherapy and mMRC score >1 point will be assigned to indacaterol maleate and glycopyrronium bromide fixed dose combination or will remain in their baseline therapy (3:1) Due to low recruitment in Groups A and B that would lead to a significant delay of trial completion, a protocol amendment was made in order to close the recruitment of Groups A and B at the time the randomization in Groups C and D would be completed. Recruitment of the Groups C and D continued as originally planned

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged ≥ 40 years
* Patients with moderate COPD according to the GOLD criteria 2013
* Current or ex-smokers who have a smoking history of at least 10 pack years
* Patients with airflow limitation indicated by a postbronchodilator FEV1 ≥50% and <80% of the predicted normal value and a post-bronchodilator FEV1/FVC <0.7 at Visit 2. Post- bronchodilator refers to within 10-15 min of inhalation of 400 μg (4x100 μg) of salbutamol
* Patients who, at Visit 1, have been for at least 3 months on a stable dose of one of the following COPD baseline treatments: *Any SABA monotherapy (such as, but not limited to, salbutamol) *Any SAMA monotherapy (such as, but not limited to, ipratropium) *Any SABA and SAMA in free or FDC (such as, but not limited to, salbutamol/ipratropium) *Any LABA monotherapy (such as, but not limited to, formoterol, salmeterol, indacaterol) *Any LAMA monotherapy (such as, but not limited to, tiotropium, aclidinium) except glycopyrronium bromide (NVA237) *Any LABA and ICS in free (ICS such as, but not limited to, beclomethasone, fluticasone) or FDC (such as, but not limited to, salmeterol/fluticasone, formoterol/budesonide).
* Patients with an mMRC score ≥1 at Visit 1.

Exclusion Criteria:

* Patients with conditions contraindicated for treatment with, or having a history of reactions/ hypersensitivity to any of the following inhaled drugs or to drugs of similar chemical classes or any component thereof: Anti-cholinergic agents, Long- and short-acting 2-adrenergic agonists, Sympathomimetic amines, Lactose or any of the other excipients of the trial medication.
* Patients with narrow-angle glaucoma or urinary retention, severe renal impairment (history of estimated glomerular filtration rate below 30 ml/min/1.73 m2 within 12 months prior to visit 1), including those with end-stage renal disease requiring dialysis.
* Patients with active/ clinical history of asthma.If the Investigator finds clear and compelling evidence that a patient was misdiagnosed with asthma in the past, then the burden of proof is on the Investigator to properly document this previous misdiagnosis. This documentation must include the rationale for this change in diagnosis including reference to the differential diagnosis that supports this decision.
* Patients with a history of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Patients who have a post-bronchodilator FEV1 decrease more than 10% compared to pre-bronchodilator FEV1 result at Visit 2 (see Appendix 5 for details).
* A documented history of >1 COPD exacerbation requiring treatment with systemic corticosteroids or antibiotics and/or hospitalization in the previous 12 months.
* Patients who have NOT had a COPD exacerbation in the previous 12 months and develop a COPD exacerbation between screening (Visit 1) and (Visit 2) will not be eligible but will be permitted to be re-screened after a minimum of 6 weeks after the resolution of the COPD exacerbation. (Patients suffering an exacerbation between Visit 1 and Visit 2 can only be re-screened in case it is the first one in the previous 12 months. In case this COPD exacerbation has led to an alteration of the patient COPD treatment, before this patient can be re-screened 3 months of stable COPD treatment will be required as described in Inclusion Criterion 6).
* Patients who, in the judgment of the investigator, have a clinically relevant laboratory abnormality or a clinically significant condition such as (but not limited to): *Unstable ischemic heart disease, left ventricular failure (NYHA Class III & IV), history of myocardial infarction,arrhythmia (excluding chronic stable atrial fibrillation). Patients with such events not considered clinically significant by the investigator may be considered for inclusion in the study.*Uncontrolled hypo-or hyperthyroidism, hypokalaemia or hyperadrenergic state. *Any condition which might compromise patient safety or compliance, interfere with evaluation, or preclude completion of the study
* History of resting QTc (Fridericia preferred, but Bazett acceptable) >450 msec (male) or >460 msec (female) within five years before Visit 1.
* Patients who are treated with glycopyrronium bromide (NVA237) at visit 1 are not allowed to be included into the trialPatients on non-selective beta-blockers. Those patients may enter the study after non-selective beta-blocker withdrawal during a 7-day wash-out period.
* Patients receiving any other prohibited COPD-related medications specified in Table 5-2 Prohibited COPD related medications must undergo the required wash-out period prior to Visit 2.
* Patients who are, in the opinion of the investigator known to be unreliable or non-compliant.
* Patients with a body mass index (BMI) of more than 40 kg/m2.
* Use of other investigational drugs within 5 half-lives of enrollment or within 30 days, whichever is longer.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study treatment.

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4389 (Actual)
Dates: Start 2014-02-14 (Actual); Primary Completion 2016-04-29 (Actual); Study Completion 2016-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (450):
- Austria (9):
  - Novartis Investigative Site, Amstetten
  - Novartis Investigative Site, Feldkirch
  - Novartis Investigative Site, Hallein
  - Novartis Investigative Site, Kirchdorf an der Krems
  - Novartis Investigative Site, Leoben
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Perg
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Wels
- Belgium (33):
  - Novartis Investigative Site, Gosselies, BEL
  - Novartis Investigative Site, Gozée, BEL
  - Novartis Investigative Site, Zichem, BEL
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Balen
  - Novartis Investigative Site, Braine-l'Alleud
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Erpent
  - Novartis Investigative Site, Éghezée
  - Novartis Investigative Site, Geraardsbergen
  - Novartis Investigative Site, Gilly
  - Novartis Investigative Site, Halen
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Heusy
  - Novartis Investigative Site, Ieper
  - Novartis Investigative Site, Knokke-Heist
  - Novartis Investigative Site, Lebbeke
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Maaseik
  - Novartis Investigative Site, Malmedy
  - Novartis Investigative Site, Mechelen
  - Novartis Investigative Site, Melsbroek
  - Novartis Investigative Site, Merksem
  - Novartis Investigative Site, Montegnée
  - Novartis Investigative Site, Natoye
  - Novartis Investigative Site, Paal-Beringen
  - Novartis Investigative Site, Ronse
  - Novartis Investigative Site, Saint-Médard
  - Novartis Investigative Site, Seraing
  - Novartis Investigative Site, Tournai
  - Novartis Investigative Site, Verviers
  - Novartis Investigative Site, Vilvoorde
  - Novartis Investigative Site, Zottegem
- Czechia (22):
  - Novartis Investigative Site, Boskovice, Czech Republic
  - Novartis Investigative Site, Brandýs nad Labem, Czech Republic
  - Novartis Investigative Site, Brno-Královo Pole, Czech Republic
  - Novartis Investigative Site, Cvikov, Czech Republic
  - Novartis Investigative Site, Havlíčkův Brod, Czech Republic
  - Novartis Investigative Site, Jirkov, Czech Republic
  - Novartis Investigative Site, Kuřim, Czech Republic
  - Novartis Investigative Site, Liberec, Czech Republic
  - Novartis Investigative Site, Lovosice, Czech Republic
  - Novartis Investigative Site, Neratovice, Czech Republic
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Pardubice, Czech Republic
  - Novartis Investigative Site, Pilsen, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Rokycany, Czech Republic
  - Novartis Investigative Site, Rudná, Czech Republic
  - Novartis Investigative Site, Teplice, Czech Republic
  - Novartis Investigative Site, Třebíč, Czech Republic
  - Novartis Investigative Site, Varnsdorf, Czech Republic
  - Novartis Investigative Site, Znojmo, Czech Republic
  - Novartis Investigative Site, Žatec, Czech Republic
  - Novartis Investigative Site, Prague
- Denmark (5):
  - Novartis Investigative Site, Alleroed
  - Novartis Investigative Site, Greve
  - Novartis Investigative Site, Haslev
  - Novartis Investigative Site, Søborg
  - Novartis Investigative Site, Værløse
- Estonia (3):
  - Novartis Investigative Site, Paide
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- France (16):
  - Novartis Investigative Site, Tours, Indre Et Loire
  - Novartis Investigative Site, Briis-sous-Forges
  - Novartis Investigative Site, Chamalières
  - Novartis Investigative Site, Châtellerault
  - Novartis Investigative Site, Forbach
  - Novartis Investigative Site, L'Aigle
  - Novartis Investigative Site, La Bouëxière
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Mûrs-Erigné
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Saint-Jean-de-Luz
  - Novartis Investigative Site, Saint-Laurent-du-Var
  - Novartis Investigative Site, Saint-Pierre
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulon
- Germany (139):
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Peine, Lower Saxony
  - Novartis Investigative Site, Koblenz, North Rhine-Westphalia
  - Novartis Investigative Site, Warendorf, North Rhine-Westphalia
  - Novartis Investigative Site, Essen, Rhineland-Palatinate
  - Novartis Investigative Site, Cottbus, Saxony
  - Novartis Investigative Site, Geesthacht, Schleswig-Holstein
  - Novartis Investigative Site, Annaberg-Buchholz
  - Novartis Investigative Site, Auerbach
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Neustadt an der Saale
  - Novartis Investigative Site, Bad Salzuflen
  - Novartis Investigative Site, Bad Wörishofen
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Bensheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Bruchsal
  - Novartis Investigative Site, Burgwedel
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Daaden
  - Novartis Investigative Site, Dachau
  - Novartis Investigative Site, Deggendorf
  - Novartis Investigative Site, Deggingen
  - Novartis Investigative Site, Delitzsch
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düren
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Eisenach
  - Novartis Investigative Site, Elsterwerda
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Föhren
  - Novartis Investigative Site, Frankenberg (Eder)
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Freudenberg
  - Novartis Investigative Site, Fürstenwalde
  - Novartis Investigative Site, Garmisch-Partenkirchen
  - Novartis Investigative Site, Gauting
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Gifhorn
  - Novartis Investigative Site, Goch
  - Novartis Investigative Site, Görlitz
  - Novartis Investigative Site, Gummersbach
  - Novartis Investigative Site, Gütersloh
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Halberstadt
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Hettstedt
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Hoyerswerda
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Jerichow
  - Novartis Investigative Site, Kamen
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Kleve
  - Novartis Investigative Site, Köthen
  - Novartis Investigative Site, Landau-Pfalz
  - Novartis Investigative Site, Landsberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Leonberg
  - Novartis Investigative Site, Leverkusen
  - Novartis Investigative Site, Limburgerhof
  - Novartis Investigative Site, Löhne
  - Novartis Investigative Site, Ludwigsburg
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Lüdenscheid
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Mayen
  - Novartis Investigative Site, Meine
  - Novartis Investigative Site, Meissen
  - Novartis Investigative Site, Menden
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Mittweida
  - Novartis Investigative Site, Mülheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münnerstadt
  - Novartis Investigative Site, Neu-Isenburg
  - Novartis Investigative Site, Neu-Ulm
  - Novartis Investigative Site, Neunkirchen
  - Novartis Investigative Site, Neuss
  - Novartis Investigative Site, Neuwied
  - Novartis Investigative Site, Northeim
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Obermichelbach
  - Novartis Investigative Site, Oschatz
  - Novartis Investigative Site, Oschersleben
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Papenburg
  - Novartis Investigative Site, Passau
  - Novartis Investigative Site, Plauen
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Prien A. Chiemsee
  - Novartis Investigative Site, Radebeul
  - Novartis Investigative Site, Ratingen
  - Novartis Investigative Site, Raubach
  - Novartis Investigative Site, Reinfeld
  - Novartis Investigative Site, Rheine
  - Novartis Investigative Site, Rodenbach
  - Novartis Investigative Site, Roth
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Rüsselsheim am Main
  - Novartis Investigative Site, Saalfeld
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Schleswig
  - Novartis Investigative Site, Schwabach
  - Novartis Investigative Site, Schwedt
  - Novartis Investigative Site, Schwerin
  - Novartis Investigative Site, Schwetzingen
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Sinsheim
  - Novartis Investigative Site, Solingen
  - Novartis Investigative Site, Sonneberg
  - Novartis Investigative Site, Strausberg
  - Novartis Investigative Site, Teuchern
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wardenburg
  - Novartis Investigative Site, Weilheim
  - Novartis Investigative Site, Welzheim
  - Novartis Investigative Site, Westerkappeln
  - Novartis Investigative Site, Wiesloch
  - Novartis Investigative Site, Wissen
  - Novartis Investigative Site, Witten
  - Novartis Investigative Site, Wolfsburg
  - Novartis Investigative Site, Wöllstein
  - Novartis Investigative Site, Zerbst
- Greece (3):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Serres
- Hungary (12):
  - Novartis Investigative Site, Győr, HUN
  - Novartis Investigative Site, Százhalombatta, HUN
  - Novartis Investigative Site, Cegléd
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Hatvan
  - Novartis Investigative Site, Komárom
  - Novartis Investigative Site, Makó
  - Novartis Investigative Site, Mátészalka
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Tatabánya
  - Novartis Investigative Site, Törökbálint
- Ireland (2):
  - Novartis Investigative Site, County Limerick
  - Novartis Investigative Site, Dublin
- Italy (47):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Avellino, AV
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Terlizzi, BA
  - Novartis Investigative Site, Triggiano, BA
  - Novartis Investigative Site, Romano di Lombardia, BG
  - Novartis Investigative Site, Feltre, BL
  - Novartis Investigative Site, Telese Terme, BN
  - Novartis Investigative Site, San Pietro Vernotico, BR
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Campobasso, CB
  - Novartis Investigative Site, Marcianise, CE
  - Novartis Investigative Site, Caltanissetta, CL
  - Novartis Investigative Site, Saluzzo, CN
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Forlì, FC
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, San Severo, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Livorno, LI
  - Novartis Investigative Site, Lodi, LO
  - Novartis Investigative Site, Lido di Camaiore, LU
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Nuoro, NU
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Piacenza, PC
  - Novartis Investigative Site, Cittadella, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pordenone, PN
  - Novartis Investigative Site, Voghera, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Riccione, RN
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Sondalo, SO
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Terni, TR
  - Novartis Investigative Site, Montebelluna, TV
  - Novartis Investigative Site, Vittorio Veneto, TV
  - Novartis Investigative Site, Busto Arsizio, VA
  - Novartis Investigative Site, Arzignano, VI
  - Novartis Investigative Site, Vicenza, VI
  - Novartis Investigative Site, Bussolengo, VR
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Torino
- Latvia (5):
  - Novartis Investigative Site, Balvi, LVA
  - Novartis Investigative Site, Jūrmala, LVA
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Riga
- Lithuania (8):
  - Novartis Investigative Site, Vilnius, LTU
  - Novartis Investigative Site, Kaunas, LT
  - Novartis Investigative Site, Vilnius, LT
  - Novartis Investigative Site, Alytus
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Utena
  - Novartis Investigative Site, Vilnius
- Norway (8):
  - Novartis Investigative Site, Førde
  - Novartis Investigative Site, Kløfta
  - Novartis Investigative Site, Lierskogen
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Skedsmokorset
  - Novartis Investigative Site, Skien
  - Novartis Investigative Site, Stavanger
  - Novartis Investigative Site, Tananger
- Poland (8):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Nowy Dwór Mazowiecki
  - Novartis Investigative Site, Ostrów Wielkopolski
  - Novartis Investigative Site, Piła
  - Novartis Investigative Site, Sopot
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (8):
  - Novartis Investigative Site, Aveiro
  - Novartis Investigative Site, Barcelos
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Guimarães
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Vila Franca de Xira
  - Novartis Investigative Site, Vila Nova de Gaia
- Romania (8):
  - Novartis Investigative Site, Bucharest, District 3
  - Novartis Investigative Site, Iași, Jud. Iasi
  - Novartis Investigative Site, Bacau
  - Novartis Investigative Site, Bragadiru
  - Novartis Investigative Site, Constanța
  - Novartis Investigative Site, Râmnicu Vâlcea
  - Novartis Investigative Site, Suceava
  - Novartis Investigative Site, Timișoara
- Russia (13):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Tomsk
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Yaroslavl
- Slovakia (12):
  - Novartis Investigative Site, Bardejov, Slovak Republic
  - Novartis Investigative Site, Bojnice, Slovak Republic
  - Novartis Investigative Site, Liptovský Hrádok, Slovak Republic
  - Novartis Investigative Site, Námestovo, Slovensko
  - Novartis Investigative Site, Kráľovský Chlmec
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Poprad
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Šaľa
  - Novartis Investigative Site, Štúrovo
  - Novartis Investigative Site, Trnava
  - Novartis Investigative Site, Vráble
- Slovenia (4):
  - Novartis Investigative Site, Golnik
  - Novartis Investigative Site, Kranj
  - Novartis Investigative Site, Maribor
  - Novartis Investigative Site, Murska Sobota
- Spain (31):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Marbella, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Mallorca, Balearic Islands
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, Centelles, Barcelona
  - Novartis Investigative Site, Mataró, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Sant Joan Despí, Barcelona
  - Novartis Investigative Site, Vic, Barcelona
  - Novartis Investigative Site, Ponferrada, Castille and León
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Canet de Mar, Catalonia
  - Novartis Investigative Site, Sant Boi de Llobregat, Catalonia
  - Novartis Investigative Site, Vic, Catalonia
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, Mérida, Extremadura
  - Novartis Investigative Site, Motril, Granada
  - Novartis Investigative Site, Valdemoro, Madrid
  - Novartis Investigative Site, Madrid, Madrid, Communidad de
  - Novartis Investigative Site, Móstoles, Madrid, Communidad de
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, Benidorm, Valencia
  - Novartis Investigative Site, Port de Sagunt, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Santiago de Compostela
  - Novartis Investigative Site, Zaragoza
- Sweden (11):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Gustavsberg
  - Novartis Investigative Site, Helsingborg
  - Novartis Investigative Site, Höllviken
  - Novartis Investigative Site, Kungshamn
  - Novartis Investigative Site, Limhamn
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Råå
  - Novartis Investigative Site, Umeå
  - Novartis Investigative Site, Västra Frölunda
  - Novartis Investigative Site, Linköping, Östergötland County
- United Kingdom (43):
  - Novartis Investigative Site, Aylesbury, Bucks
  - Novartis Investigative Site, Fowey, Cornwall
  - Novartis Investigative Site, Liskeard, Cornwall
  - Novartis Investigative Site, Penzance, Cornwall
  - Novartis Investigative Site, Redruth, Cornwall
  - Novartis Investigative Site, St Austell, Cornwall
  - Novartis Investigative Site, Torpoint, Cornwall
  - Novartis Investigative Site, Bath, England
  - Novartis Investigative Site, Havant, Hampshire
  - Novartis Investigative Site, Burbage, Leicester
  - Novartis Investigative Site, Daventry, Northamptonshire
  - Novartis Investigative Site, Sneinton, Nottingham
  - Novartis Investigative Site, Axbridge, Somerset
  - Novartis Investigative Site, Frome, Somerset
  - Novartis Investigative Site, Taunton, Somerset
  - Novartis Investigative Site, South Shields, Tyne and Wear
  - Novartis Investigative Site, Barry, Vale Of Glamorgan
  - Novartis Investigative Site, Royal Leamington Spa, Warwickshire
  - Novartis Investigative Site, Crawley, West Sussex
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Trowbridge, Wiltshire
  - Novartis Investigative Site, Strensall, Yorkshire
  - Novartis Investigative Site, Bexhill-on-Sea
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Chadderton
  - Novartis Investigative Site, Cheshire
  - Novartis Investigative Site, Chesterfield
  - Novartis Investigative Site, Chippenham
  - Novartis Investigative Site, Coventry
  - Novartis Investigative Site, Hamilton
  - Novartis Investigative Site, Lancashire
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Motherwell
  - Novartis Investigative Site, Oldham
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Shrewsbury
  - Novartis Investigative Site, South Yorkshire
  - Novartis Investigative Site, Stockton-on-Tees
  - Novartis Investigative Site, Vale of Glanmorgan
  - Novartis Investigative Site, Watford
  - Novartis Investigative Site, Wiltshire
  - Novartis Investigative Site, Wishaw

REFERENCES:
- [Derived] Greulich T, Kostikas K, Gaga M, Aalamian-Mattheis M, Lossi NS, Patalano F, Nunez X, Pagano VA, Fogel R, Vogelmeier CF, Clemens A. Indacaterol/glycopyrronium reduces the risk of clinically important deterioration after direct switch from baseline therapies in patients with moderate COPD: a post hoc analysis of the CRYSTAL study. Int J Chron Obstruct Pulmon Dis. 2018 Apr 16;13:1229-1237. doi: 10.2147/COPD.S159732. eCollection 2018. PMID 29713156
- [Derived] Vogelmeier CF, Gaga M, Aalamian-Mattheis M, Greulich T, Marin JM, Castellani W, Ninane V, Lane S, Nunez X, Patalano F, Clemens A, Kostikas K; CRYSTAL study investigators. Efficacy and safety of direct switch to indacaterol/glycopyrronium in patients with moderate COPD: the CRYSTAL open-label randomised trial. Respir Res. 2017 Jul 18;18(1):140. doi: 10.1186/s12931-017-0622-x. PMID 28720132

RESULTS

PARTICIPANT FLOW:
Groups:
- A1 (Any SABA and/or SAMA): Patients treated with any SABA and/or SAMA as monotherapy or in free or fixed dose combination at enrollment and randomized to remain in their baseline therapy with any SABA and/or SAMA
Period: Overall Study
Arm/Group | A1 (Any SABA and/or SAMA) | A2 (Glycopyrronium) | B1 (Any LAMA or LABA and mMRC=1) | B2 (Glycopyrronium and mMRC=1) | C1 (Any LABA and ICS) | C2 (Indacaterol/Glycopyrronium) | D1 (Any LAMA or LABA and mMRC>1) | D2 (Indacaterol/Glycopyrronium and mMRC>1)
Started | 130 | 387 | 420 | 1262 | 274 | 822 | 274 | 820
The Intention-to-treat (ITT) Population | 122 | 369 | 420 | 1254 | 269 | 811 | 268 | 811
Completed | 107 | 303 | 367 | 1033 | 234 | 666 | 237 | 699
Not Completed | 23 | 84 | 53 | 229 | 40 | 156 | 37 | 121
Not completed — Administrative problems | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 3
Not completed — Death | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 2
Not completed — Worsening of disease | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1
Not completed — Other | 2 | 9 | 7 | 17 | 4 | 8 | 4 | 7
Not completed — Protocol deviation | 6 | 31 | 25 | 84 | 17 | 47 | 15 | 42
Not completed — Moderate / severe COPD exacerbation | 5 | 14 | 12 | 40 | 6 | 40 | 8 | 19
Not completed — Subject withdrawal of consent | 3 | 6 | 2 | 28 | 4 | 19 | 0 | 20
Not completed — Adverse Event | 0 | 8 | 2 | 26 | 3 | 18 | 3 | 15
Not completed — Other | 4 | 2 | 3 | 10 | 1 | 6 | 2 | 2
Not completed — Medication non-compliance | 0 | 4 | 1 | 6 | 2 | 3 | 1 | 3
Not completed — Use of prohibited treatment | 1 | 4 | 1 | 2 | 1 | 6 | 2 | 0
Not completed — Investigator decision | 0 | 3 | 0 | 7 | 1 | 1 | 0 | 4
Not completed — Lost to Follow-up | 0 | 2 | 0 | 3 | 1 | 4 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A1 (Any SABA and/or SAMA) | A2 (Glycopyrronium) | B1 (Any LAMA or LABA and mMRC=1) | B2 (Glycopyrronium and mMRC=1) | C1 (Any LABA and ICS) | C2 (Indacaterol/Glycopyrronium) | D1 (Any LAMA or LABA and mMRC>1) | D2 (Indacaterol/Glycopyrronium and mMRC>1) | Total
Number analyzed (Participants) | 130 | 387 | 420 | 1262 | 274 | 822 | 274 | 820 | 4389
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (8.2) | 63.2 (8.3) | 64.6 (8.1) | 64.4 (8.2) | 64.4 (9.0) | 64.7 (8.7) | 65.1 (7.6) | 65.4 (8.3) | 64.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 119 | 131 | 376 | 106 | 286 | 95 | 276 | 1437
  Male | 82 | 268 | 289 | 886 | 168 | 536 | 179 | 544 | 2952

OUTCOME MEASURES:

1. Primary Outcome: Trough FEV1 at Week 12 for Group: Glycopyrronium vs. Short-acting Bronchodilators (SABA and/or SAMA as Monotherapy or in Free or FDC)
Description: Trough FEV1 at visit 4 is defined as FEV1, computed as the mean of forced expiratory volume in 1 second 15min and 45 min pre dose measurements, at the end of the dosing interval
Time Frame: Week 12 (Visit 4)
Population: The intention-to-treat (ITT) population consisted of all randomized patients who received at least one dose of the study treatment and who were getting the appropriate medication, be it glycopyrronium, indacaterol + glycopyrronium or comparative treatment (baseline therapy) in the respective comparisons of the different groups
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | A1 (Any SABA and/or SAMA) | A2 (Glycopyrronium)
Number analyzed (Participants) | 122 | 369
Liters | 1.8264 [1.7797 to 1.8732] | 1.8916 [1.8647 to 1.9185]
Statistical Analysis 1: Comparison: A1 (Any SABA and/or SAMA) vs A2 (Glycopyrronium); Test type: Superiority or Other; p = 0.0180, linear mixed model

2. Primary Outcome: Trough FEV1 at Week 12 for Group: Glycopyrronium vs. Long-acting Bronchodilators (LABA or LAMA Monotherapy)
Description: as for outcome 1
Time Frame: Week 12 (Visit 4)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | B1 (Any LAMA or LABA and mMRC=1) | B2 (Glycopyrronium and mMRC=1)
Number analyzed (Participants) | 420 | 1254
Liters | 1.8004 [1.7768 to 1.8239] | 1.8215 [1.8078 to 1.8352]
Statistical Analysis 1: Comparison: B1 (Any LAMA or LABA and mMRC=1) vs B2 (Glycopyrronium and mMRC=1); Test type: Non-Inferiority or Equivalence — H0: Glycopyrronium (50 μg o.d.) [randomized group B2] was inferior to LABA or LAMA (random group B1) with respect to mean trough FEV1 after 12 weeks of treatment. H0: μFEV1, NVA237 - μFEV1, LABA and/or LAMA < -40 mL Ha: Glycopyrronium (50 μg o.d.) [randomized group B2] is non-inferior to LABA or LAMA (random group B1) with respect to mean trough FEV1 after 12 weeks of treatment. Ha: μFEV1, NVA237 - μFEV1, LABA and/or LAMA ≥ -40 mL; p < 0.0001, linear mixed model

3. Primary Outcome: Trough FEV1 at Week 12 for Group: Indacaterol Maleate and Glycopyrronium Bromide FDC vs. LABA and ICS in Free or FDC
Description: as for outcome 1
Time Frame: Week 12 (Visit 4)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | C1 (Any LABA and ICS) | C2 (Indacaterol/Glycopyrronium)
Number analyzed (Participants) | 269 | 811
Liters | 1.6847 [1.6542 to 1.7153] | 1.7558 [1.7378 to 1.7737]
Statistical Analysis 1: Comparison: C1 (Any LABA and ICS) vs C2 (Indacaterol/Glycopyrronium); Test type: Superiority or Other; p < 0.0001, linear mixed model

4. Primary Outcome: Trough FEV1 at Week 12 for Group: Indacaterol Maleate and Glycopyrronium Bromide FDC vs. Long-acting Bronchodilators (LABA or LAMA Monotherapy)
Description: as for outcome 1
Time Frame: Week 12 (Visit 4)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | D1 (Any LAMA or LABA and mMRC>1) | D2 (Indacaterol/Glycopyrronium and mMRC>1)
Number analyzed (Participants) | 268 | 811
Liters | 1.6728 [1.6461 to 1.6994] | 1.7742 [1.7587 to 1.7896]
Statistical Analysis 1: Comparison: D1 (Any LAMA or LABA and mMRC>1) vs D2 (Indacaterol/Glycopyrronium and mMRC>1); Test type: Superiority or Other; p < 0.0001, linear mixed model

5. Primary Outcome: Change From Baseline on Transition Dyspnea Index (TDI) for Groups: Glycopyrronium vs. Short-acting Bronchodilators (SABA and/or SAMA as Monotherapy or in Free or FDC)
Description: Transition Dyspnea Index (TDI) captures changes from baseline. The TDI score is based on three domains with each domain scored from -3 (major deterioration) to +3 (major improvement), to give an overall score of -9 to +9, a negative score indicating a deterioration from baseline. A TDI focal score of 1 is considered to be a clinically significant improvement from baseline.
Time Frame: Day 1 (baseline) and week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | A1 (Any SABA and/or SAMA) | A2 (Glycopyrronium)
Number analyzed (Participants) | 122 | 369
Units on a scale | 0.5117 [-0.0073 to 1.0306] | 2.3005 [2.0015 to 2.5995]
Statistical Analysis 1: Comparison: A1 (Any SABA and/or SAMA) vs A2 (Glycopyrronium); Test type: Superiority or Other; p < 0.0001, linear mixed model

6. Primary Outcome: Change From Baseline on Transition Dyspnea Index (TDI) for Groups: Glycopyrronium vs. Long-acting Bronchodilators (LABA or LAMA Monotherapy)
Description: as for outcome 5
Time Frame: Day 1 (baseline) and week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | B1 (Any LAMA or LABA and mMRC=1) | B2 (Glycopyrronium and mMRC=1)
Number analyzed (Participants) | 420 | 1254
Units on a scale | 0.6969 [0.4169 to 0.9769] | 1.4351 [1.2718 to 1.5984]
Statistical Analysis 1: Comparison: B1 (Any LAMA or LABA and mMRC=1) vs B2 (Glycopyrronium and mMRC=1); Test type: Non-Inferiority or Equivalence — A difference of 0.6 points in TDI was adopted as boundary for non-inferiority; p < 0.0001, linear mixed model

7. Primary Outcome: Change From Baseline on Transition Dyspnea Index (TDI) for Groups: Indacaterol Maleate and Glycopyrronium Bromide FDC vs. LABA and ICS in Free or FDC
Description: as for outcome 5
Time Frame: Day 1 (baseline) and week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | C1 (Any LABA and ICS) | C2 (Indacaterol/Glycopyrronium)
Number analyzed (Participants) | 269 | 811
Units on a scale | 0.8508 [0.4676 to 1.2340] | 1.9491 [1.7207 to 2.1775]
Statistical Analysis 1: Comparison: C1 (Any LABA and ICS) vs C2 (Indacaterol/Glycopyrronium); Test type: Superiority or Other; p < 0.0001, linear mixed model

8. Primary Outcome: Change From Baseline on Transition Dyspnea Index (TDI) for Groups: Indacaterol Maleate and Glycopyrronium Bromide FDC vs. Long-acting Bronchodilators (LABA or LAMA Monotherapy)
Description: as for outcome 5
Time Frame: Day 1 (baseline) and week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | D1 (Any LAMA or LABA and mMRC>1) | D2 (Indacaterol/Glycopyrronium and mMRC>1)
Number analyzed (Participants) | 268 | 811
Units on a scale | 0.8632 [0.5098 to 1.2166] | 2.1209 [1.9130 to 2.3288]
Statistical Analysis 1: Comparison: D1 (Any LAMA or LABA and mMRC>1) vs D2 (Indacaterol/Glycopyrronium and mMRC>1); Test type: Superiority or Other; p < 0.0001, linear mixed model

9. Secondary Outcome: Trough FEV1 at Week 12 for Group: Glycopyrronium vs. Short-acting Bronchodilators (SABA and/or SAMA as Monotherapy or in Free or FDC) or vs. Long-acting Bronchodilators (LABA or LAMA Monotherapy)
Description: as for outcome 1
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- A2 + B2: A2 (glycopyrronium)+B2 (glycopyrronium and mMRC=1
- A1 + B1: A1(any SABA and/or SAMA+B1 (any LAMA or LABA and mMRC=1
Arm/Group | A2 + B2 | A1 + B1
Number analyzed (Participants) | 1623 | 542
Liters | 1.8373 [1.8250 to 1.8496] | 1.8065 [1.7853 to 1.8276]

10. Secondary Outcome: Change From Baseline on on Transition Dyspnea Index (TDI) for Groups: Glycopyrronium vs. Short-acting Bronchodilators (SABA and/or SAMA as Monotherapy or in Free or FDC) or Long-acting Bronchodilators (LABA or LAMA Monotherapy)
Description: as for outcome 5
Time Frame: Day 1 (baseline) and week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- A2 +B2: A2 (glycopyrronium)+B2 (glycopyrronium and mMRC=1
- A1 +B1: A1(any SABA and/or SAMA+B1 (any LAMA or LABA and mMRC=1)
Arm/Group | A2 +B2 | A1 +B1
Number analyzed (Participants) | 1623 | 542
Score on a scale | 1.6315 [1.4874 to 1.7756] | 0.6562 [0.4085 to 0.9039]

11. Secondary Outcome: Trough FEV1 at Week 12 for Group: Indacaterol Maleate and Glycopyrronium Bromide FDC vs. LABA or LAMA Monotherapy or LABA and ICS in Free or FDC on Trough FEV1 at Week 12.
Description: as for outcome 1
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- C2 +D2: C2 (indacaterol/glycopyrronium)+D2 (indacaterol/glycopyrronium and mMRC>1)
- C1 + D1: C1 (any LABA and ICS)+D1 (any LAMA or LABA and mMRC>1)
Arm/Group | C2 +D2 | C1 + D1
Number analyzed (Participants) | 1622 | 537
Liters | 1.7650 [1.7532 to 1.7768] | 1.6789 [1.6587 to 1.6992]

12. Secondary Outcome: Change From Baseline on Transition Dyspnea Index (TDI) for Groups: Indacaterol Maleate and Glycopyrronium Bromide FDC vs. LABA or LAMA Monotherapy or LABA and ICS in Free or FDC
Description: as for outcome 5
Time Frame: Day 1 (baseline) and week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- C2 +D2: C2 (indacaterol/glycopyrronium) + D2 (indacaterol/glycopyrronium and mMRC>1)
- C1 + D1: C1 (any LABA and ICS) + D1 (any LAMA or LABA and mMRC>1)
Arm/Group | C2 +D2 | C1 + D1
Number analyzed (Participants) | 1622 | 537
Score on a scale | 2.0354 [1.8811 to 2.1896] | 0.8588 [0.5983 to 1.1192]

13. Secondary Outcome: Change From Baseline on Total Score of COPD Assessment Test (CAT) for Groups: Glycopyrronium and Indacaterol Maleate and Glycopyrronium Bromide FDC
Description: Total score of COPD Assessment Test (CAT) will be measured at baseline and at week 12. This questionnaire is completed by the patient. The score ranges from 0-40 where higher scores represent worse health status. CAT scores ≥ 10 are associated with significantly impaired health status.
Time Frame: Day 1 (baseline) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | A1 (Any SABA and/or SAMA) | A2 (Glycopyrronium) | B1 (Any LAMA or LABA and mMRC=1) | B2 (Glycopyrronium and mMRC=1) | C1 (Any LABA and ICS) | C2 (Indacaterol/Glycopyrronium) | D1 (Any LAMA or LABA and mMRC>1) | D2 (Indacaterol/Glycopyrronium and mMRC>1)
Number analyzed (Participants) | 122 | 369 | 420 | 1254 | 269 | 811 | 268 | 811
Score | 0.1 (4.6) | -1.8 (5.3) | 0.1 (4.9) | -0.5 (4.6) | -0.4 (4.8) | -1.4 (5.4) | -0.9 (5.0) | -1.9 (5.3)

14. Secondary Outcome: Change From Baseline on Total Score of Clinical COPD Questionnaire (CCQ) for Groups: Glycopyrronium and Indacaterol Maleate and Glycopyrronium Bromide FDC
Description: The Clinical COPD Questionnaire (CCQ) is a self-administered 10-item questionnaire developed to measure clinical control in patients with COPD. Patients will be instructed to recall their experiences during the previous week. They respond to each question using a 7-point scale from 0 = asymptomatic/no imitation to 6 = extremely symptomatic/totally limited. The questionnaire is divided into 3 domains (symptoms [items 1, 2, 5, and 6] functional [items 7, 8, 9, and 10] and mental state [items 3 and 4]). The overall clinical COPD control score and the scores of the domains are calculated by adding all the scores together and dividing this sum by the number of questions.
  Thus, the overall clinical COPD control score as well as the score on each of the three domains varies between 0 (very good control) to 6 (extremely poor control).
Time Frame: Day 1 (baseline) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | A1 (Any SABA and/or SAMA) | A2 (Glycopyrronium) | B1 (Any LAMA or LABA and mMRC=1) | B2 (Glycopyrronium and mMRC=1) | C1 (Any LABA and ICS) | C2 (Indacaterol/Glycopyrronium) | D1 (Any LAMA or LABA and mMRC>1) | D2 (Indacaterol/Glycopyrronium and mMRC>1)
Number analyzed (Participants) | 122 | 369 | 420 | 1254 | 269 | 811 | 268 | 811
Score | -0.0 (0.6) | -0.3 (0.7) | 0.0 (0.7) | -0.1 (0.7) | -0.1 (0.7) | -0.2 (0.8) | -0.1 (0.8) | -0.3 (0.8)

15. Secondary Outcome: Mean Number of Puffs of Rescue Medication Use for Groups: Glycopyrronium and Indacaterol Maleate and Glycopyrronium Bromide FDC
Description: Mean number of puffs of rescue medication use will be measured using eDiary data over 12 weeks of treatment.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of puffs
Arm/Group | A1 (Any SABA and/or SAMA) | A2 (Glycopyrronium) | B1 (Any LAMA or LABA and mMRC=1) | B2 (Glycopyrronium and mMRC=1) | C1 (Any LABA and ICS) | C2 (Indacaterol/Glycopyrronium) | D1 (Any LAMA or LABA and mMRC>1) | D2 (Indacaterol/Glycopyrronium and mMRC>1)
Number analyzed (Participants) | 122 | 369 | 420 | 1254 | 269 | 811 | 268 | 811
Number of puffs | 1.8 (1.7) | 1.0 (1.3) | 0.8 (1.2) | 0.7 (1.1) | 1.6 (1.7) | 1.1 (1.4) | 1.4 (1.4) | 1.1 (1.3)

16. Secondary Outcome: Mean Change From Baseline Reported Symptoms of COPD for Groups: Glycopyrronium and Indacaterol Maleate and Glycopyrronium Bromide FDC
Description: Patient-reported symptoms of COPD combined will be measured using eDiary data reported over the 12 week treatment period. The mean total symptom scores and mean individual symptom scores for the patient were calculated for the whole study period. The mean change from baseline in the total scores and in the individual scores were summarized by treatment and were analyzed for the percentage of nights with no nighttime awakenings and percentage of days with no symptoms.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | A1 (Any SABA and/or SAMA) | A2 (Glycopyrronium) | B1 (Any LAMA or LABA and mMRC=1) | B2 (Glycopyrronium and mMRC=1) | C1 (Any LABA and ICS) | C2 (Indacaterol/Glycopyrronium) | D1 (Any LAMA or LABA and mMRC>1) | D2 (Indacaterol/Glycopyrronium and mMRC>1)
Number analyzed (Participants) | 122 | 369 | 420 | 1254 | 269 | 811 | 268 | 811
Percentage of days | -0.04 (0.15) | -0.10 (0.22) | -0.03 (0.19) | -0.05 (0.20) | -0.05 (0.19) | -0.07 (0.22) | -0.04 (0.19) | -0.09 (0.21)

ADVERSE EVENTS:
Groups:
- B1 (Any LAMA or@ LABA and mMRC eq 1): Patients treated with any LABA or LAMA monotherapy and mMRC score =1 point at Visit 1 and randomized to remain in their baseline treatment with LABA or LAMA
- B2 (Glycopyrronium@ and mMRC eq 1): Patients treated with any LABA or LAMA monotherapy and mMRC score =1 point at Visit 1 and randomized to switch in treatment with glycopyrronium (50 μg o.d.)
- C2 (Indacaterol/@Glycopyrronium): Patients treated with any LABA and ICS in free or FDC at enrollment and randomized to switch in treatment with indacaterol maleate and glycopyrronium bromide FDC (110/50 μg o.d.)
- D1 (Any LAMA or@ LABA and mMRC gt 1): Patients treated with any LABA or LAMA monotherapy and mMRC score >1 point at Visit 1 and randomized to remain their baseline in treatment with LABA or LAMA
- D2 (Indacaterol/@Glycopyrronium and@ mMRC gt 1): Patients treated with any LABA or LAMA monotherapy and mMRC score >1 point at Visit 1 and randomized to switch in treatment with indacaterol maleate and glycopyrronium bromide FDC (110/50 μg o.d.).
Arm/Group | A1 (Any SABA and/or SAMA) | A2 (Glycopyrronium) | B1 (Any LAMA or@ LABA and mMRC eq 1) | B2 (Glycopyrronium@ and mMRC eq 1) | C1 (Any LABA and ICS) | C2 (Indacaterol/@Glycopyrronium) | D1 (Any LAMA or@ LABA and mMRC gt 1) | D2 (Indacaterol/@Glycopyrronium and@ mMRC gt 1)
Serious Adverse Events (participants affected / at risk) | 4/125 | 9/385 | 11/417 | 30/1248 | 6/269 | 22/816 | 10/269 | 34/814
Other Adverse Events (participants affected / at risk) | 19/125 | 67/385 | 63/417 | 163/1248 | 29/269 | 119/816 | 20/269 | 120/814
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A1 (Any SABA and/or SAMA) (N=125) | A2 (Glycopyrronium) (N=385) | B1 (Any LAMA or@ LABA and mMRC eq 1) (N=417) | B2 (Glycopyrronium@ and mMRC eq 1) (N=1248) | C1 (Any LABA and ICS) (N=269) | C2 (Indacaterol/@Glycopyrronium) (N=816) | D1 (Any LAMA or@ LABA and mMRC gt 1) (N=269) | D2 (Indacaterol/@Glycopyrronium and@ mMRC gt 1) (N=814)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Congenital central nervous system anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diverticulum oesophageal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hernia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ulcer (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Biliary tract disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mediastinal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 7
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bursa injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Heart rate decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular dementia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 1 | 3 | 1 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Femoral artery aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ischaemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A1 (Any SABA and/or SAMA) (N=125) | A2 (Glycopyrronium) (N=385) | B1 (Any LAMA or@ LABA and mMRC eq 1) (N=417) | B2 (Glycopyrronium@ and mMRC eq 1) (N=1248) | C1 (Any LABA and ICS) (N=269) | C2 (Indacaterol/@Glycopyrronium) (N=816) | D1 (Any LAMA or@ LABA and mMRC gt 1) (N=269) | D2 (Indacaterol/@Glycopyrronium and@ mMRC gt 1) (N=814)
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1 | 3 | 0 | 2 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 4 | 4 | 4 | 1 | 1 | 1 | 3
Nasopharyngitis (Infections and infestations) | 8 | 38 | 24 | 71 | 11 | 37 | 10 | 54
Pharyngitis (Infections and infestations) | 3 | 1 | 0 | 7 | 0 | 3 | 1 | 5
Rhinitis (Infections and infestations) | 0 | 1 | 7 | 12 | 2 | 5 | 1 | 10
Tracheitis (Infections and infestations) | 2 | 0 | 2 | 2 | 0 | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 2 | 1 | 5 | 0 | 1 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6 | 3 | 8 | 2 | 10 | 2 | 11
Headache (Nervous system disorders) | 0 | 7 | 3 | 9 | 1 | 12 | 1 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 13 | 33 | 5 | 44 | 4 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 6 | 13 | 6 | 7 | 2 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 3 | 10 | 4 | 3 | 1 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 1 | 0 | 2 | 2 | 0
Hypertension (Vascular disorders) | 1 | 3 | 7 | 7 | 2 | 5 | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.